CLINICAL TRIAL: NCT05881278
Title: PRESERVE Heart Study: A Prospective, Multi-center, Single-Arm, Open-Label Study of Hearts Transplanted After Non-Ischemic Heart PRESERVation From Extended Donors
Brief Title: XVIVO Heart Perfusion System (XHPS) With Supplemented XVIVO Heart Solution (SXHS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIHP - 001
Record Dates: First submitted 2023-05-18; First posted 2023-05-31 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Transplant; Failure, Heart
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects requiring a Heart Transplant (Experimental): Device: Preservation of hearts for transplant.
  Interventions: Device: Non-Ischemic Heart Preservation (NIHP) using the XVIVO Heart Preservation System (XHPS)

INTERVENTIONS:
Device: Non-Ischemic Heart Preservation (NIHP) using the XVIVO Heart Preservation System (XHPS) — Study donor hearts meeting extended criteria are preserved via Non-Ischemic Heart Preservation (NIHP) using the XVIVO Heart Preservation System (XHPS)

SUMMARY:
The purpose of this study is to evaluate if Non-Ischemic Heart Preservation (NIHP) of extended criteria donor hearts using the XVIVO Heart Preservation System (XHPS) is a safe and effective way to preserve and transport hearts for transplantation.

DETAILED DESCRIPTION:
PRESERVE Heart Study - This is a prospective, multicenter, non-randomized, single arm, open label study in subjects requiring a Heart Transplant. Study donor hearts meeting extended criteria are preserved via Non-Ischemic Heart Preservation (NIHP) using the XVIVO Heart Preservation System (XHPS).

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Age ≥18 years.
2. Signed informed consent form (ICF).
3. Listed for heart transplantation

Recipient Exclusion Criteria:

1. Previous solid organ or bone marrow transplantation.
2. Requires a multi-organ transplant.
3. Subject is enrolled and ongoing in another investigational pharmaceutical or medical device clinical trial (Exception: observational studies are permitted).
4. Subject is on mechanical circulatory support pre-transplant other than durable LVAD, Impella or intra-aortic balloon pump.
5. History of complex congenital heart disease ie: single ventricle physiology (Per Investigators discretion).
6. Subject on renal replacement therapy/dialysis.
7. Ventilator dependence (subject is intubated at time of transplant/unable to provide consent or re-affirmation of consent).
8. Sensitized subject is undergoing desensitization treatment.

Donor Inclusion Criteria:

1. Estimated Cross Clamp Time ≥ 4 hours, OR
2. Estimated Cross Clamp Time ≥ 2 hours, AND

   Any ONE or more of the following:
   * Age ≥ 50 years
   * LVEF 40-50% at time of provisional acceptance
   * Down-time ≥ 20 mins
   * Hypertrophy/Septal thickness >12- ≤16mm
   * Angiographic luminal irregularities with no significant CAD, OR
3. Donation after Circulatory Death (DCD) donors.

Donor Exclusion Criteria:

1. Unstable hemodynamics requiring high-dose inotropic support.
2. Significantly abnormal coronary angiogram defined as CAD > 50% stenosis of one or more vessels.
3. Moderate to severe cardiac valve pathology.
4. Investigator's clinical decision to exclude from trial.
5. Previous Sternotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of patient survival | Post-operative Day 365.
  The percentage of patient survival at 365 days from the date of transplant. The long-term safety success is defined as survival.
The percentage of patient treatment success rate | 30 days post transplantation
  The percentage of patient treatment success rate at 30-days post transplantation. The treatment success is defined as freedom from treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Tiwari, Study Director — XVIVO Perfusion
Locations (20):
- United States (20):
  - University of California San Diego, La Jolla, California
  - Cedars-Sinai, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford Medicine, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Maryland Medical Center/University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No